CLINICAL TRIAL: NCT02776345
Title: Study to Evaluate Ultrasound Guided Interventions of Calcific Tendonitis of Rotator Cuff- International CollabratioN (SUCTION)
Brief Title: Ultrasound Guided Interventions of Calcific Tendonitis of Rotator Cuff (SUCTION)
Acronym: SUCTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Hema Choudur, Associate Professor, Department of Radiology, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1447
Record Dates: First submitted 2016-04-15; First posted 2016-05-18 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Rotator Cuff Calcific Tendonitis
Keywords: calcific tendonitis; rotator cuff calcific tendonitis
MeSH Terms: interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasound guided Needle Fragmentation (Active Comparator): Ultrasound guided Needle Fragmentation (Intervention):
  Using 15-20 to and fro gentle movements of the needle tip, the calcification will be fragmented, with the needle tip within the pseudocapsule. The needle tip will be retracted into the subacromial bursa and 3 ml of 0.5% sensorcaine and 1 ml of steroid ( Depomedrol- 40mg/ml) will be injected into the bursa. The needle will then be removed.
  Interventions: Other: Ultrasound guided Needle Fragmentation
- US guided needle fragmentation & Lavage (Active Comparator): Using local anesthetic and strict aseptic precautions, the tip of the 18-20 gauge needle will be advanced into the sub acromial bursa under ultrasound guidance and 2ml. of local anesthetic ( 1% xylocaine) will be injected into the bursa. The needle tip will be advanced into the supraspinatus tendon and ½ ml or less of 0.5% Sensorcaine will be injected into the pseudo capsule around the calcification. Using 15-20 to and fro gentle movements of the needle tip, the calcification will be fragmented, with the needle tip within the pseudo capsule. During this procedure, or after the fragmentation, using a syringe of saline or local anesthetic( 1% xylocaine) and with pumping action of the syringe the calcification with be sucked into the syringe.
  Interventions: Other: US guided needle fragmentation & Lavage
- Ultrasound guided subacromial injection (Placebo Comparator): Using local anesthetic and strict aseptic precautions, the tip of the 22 gauge needle will be advanced into the sub acromial bursa under ultrasound guidance and 4 ml. of local anesthetic ( 0.5% xylocaine) and 1 ml of steroid( Depomedrol 40 mg/ml) will be injected into the bursa. The needle will then be removed. Post procedure US images in the short and long axis planes will be obtained and documented. The patient's post procedure pain on a scale of 10 and their range of shoulder movement (abduction) will be assessed and documented.
  Interventions: Other: Ultrasound guided subacromial injection

INTERVENTIONS:
Other: Ultrasound guided Needle Fragmentation — Using 15-20 to and fro gentle movements of the needle tip, the calcification will be fragmented, with the needle tip within the pseudocapsule. The needle tip will be retracted into the subacromial bursa and 3 ml of 0.5% sensorcaine and 1 ml of steroid ( Depomedrol- 40mg/ml) will be injected into the bursa. The needle will then be removed.
  Arms: Ultrasound guided Needle Fragmentation
Other: US guided needle fragmentation & Lavage — Using local anesthetic and strict aseptic precautions, the tip of the 18-20 gauge needle will be advanced into the sub acromial bursa under ultrasound guidance and 2ml. of local anesthetic ( 1% xylocaine) will be injected into the bursa. The needle tip will be advanced into the supraspinatus tendon and ½ ml or less of 0.5% Sensorcaine will be injected into the pseudo capsule around the calcification. Using 15-20 to and fro gentle movements of the needle tip, the calcification will be fragmented, with the needle tip within the pseudo capsule. During this procedure, or after the fragmentation, using a syringe of saline or local anesthetic( 1% xylocaine) and with pumping action of the syringe the calcification with be sucked into the syringe.
  Arms: US guided needle fragmentation & Lavage
Other: Ultrasound guided subacromial injection — Using local anesthetic and strict aseptic precautions, the tip of the 22 gauge needle will be advanced into the sub acromial bursa under ultrasound guidance and 4 ml. of local anesthetic ( 0.5% xylocaine) and 1 ml of steroid( Depomedrol 40 mg/ml) will be injected into the bursa. The needle will then be removed. Post procedure US images in the short and long axis planes will be obtained and documented. The patient's post procedure pain on a scale of 10 and their range of shoulder movement (abduction) will be assessed and documented.
  Arms: Ultrasound guided subacromial injection

SUMMARY:
The purpose of this study is to determine whether minimally invasive treatments like ultrasound guided needle fragmentation with and without lavage is associated with better clinical outcomes compared to the subacromial bursal corticosteroid injection treatment only.

DETAILED DESCRIPTION:
The objectives of this study are to compare the clinical outcomes of the three treatment arms: ultrasound guided needle fragmentation with lavage, ultrasound guided needle fragmentation without lavage, and subacromial bursal corticosteroid injection treatment. The study design is a randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women ages 18 to 60 years
2. Shoulder pain ( including impingement pain) and reduced range of shoulder movement for greater than 6 months with no relief from non-operative means (physiotherapy, nonsteroidal anti-inflammatory medication, rest).
3. Documentation of failed physiotherapy and conservative management.
4. Calcific tendonitis as diagnosed on ultrasound.
5. Informed consent from participant.
6. Ability to speak, understand and read in the language of the clinical site.

Exclusion Criteria:

1. Previous inclusion in a study involving calcific tendonitis of the rotator cuff
2. Evidence of a calcification in any of the rotator cuff tendons except the supraspinatus tendon.
3. Presence of a tear of the rotator cuff.
4. The supraspinatus tendon calcification is more than 1.5 cm is its largest dimension.
5. Concomitant clinical or MRI diagnosis of frozen shoulder.
6. Previous rotator cuff or shoulder surgery.
7. Those on blood thinners.
8. Those with allergies to medication used.
9. Those with a skin infection at the site of needle entry.
10. Immunosuppressive medication use.
11. Chronic pain syndromes.
12. Significant medical co-morbidities (requiring daily assistance).
13. Ongoing litigation or compensation claims secondary to shoulder problems.
14. Age below 18 years and above 60 years.
15. Any other reasons given to exclude the patient.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Decrease in Pain as measured by the Visual analog scale from 1-10 | 8 months
  Pain in the original symptomatic area of the rotator cuff will be reassessed using the visual analog scale from 1-10 (1 being the lowest pain and 10 being the highest)
Decreased Range of Motion in the shoulder measured in degrees | 8 months
  Abduction, internal rotation, external rotation and circumduction of the shoulder

SECONDARY OUTCOMES:
Complications and co existing conditions not detected prior to the procedure | Post ultrasound guided procedure through completion of study, up to one year
  Infection, procedure induced tendon tears, reduced range of motion ( from other causes such as frozen shoulder), and other adverse events
Costs and health resource utilization as measured by administrative and billing data related to treatment | Up to 8-12 months post surgery
  Treatment-related costs to the healthcare system and/or patient through billing codes and data
Generic physical and mental health as measured by EuroQol | Up to 8-12 months post surgery
The ultrasound appearance of the targeted calcification | Up to 8-12 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hema N Choudur, MBBS, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fusaro I, Orsini S, Diani S, Saffioti G, Zaccarelli L, Galletti S. Functional results in calcific tendinitis of the shoulder treated with rehabilitation after ultrasonic-guided approach. Musculoskelet Surg. 2011 Jul;95 Suppl 1:S31-6. doi: 10.1007/s12306-011-0119-6. PMID 21479869
- [Background] Kachewar SG, Kulkarni DS. Calcific tendinitis of the rotator cuff: a review. J Clin Diagn Res. 2013 Jul;7(7):1482-5. doi: 10.7860/JCDR/2013/4473.3180. Epub 2013 Jul 1. PMID 23998102
- [Background] del Cura JL, Torre I, Zabala R, Legorburu A. Sonographically guided percutaneous needle lavage in calcific tendinitis of the shoulder: short- and long-term results. AJR Am J Roentgenol. 2007 Sep;189(3):W128-34. doi: 10.2214/AJR.07.2254. PMID 17715078
- [Background] Yoo JC, Koh KH, Park WH, Park JC, Kim SM, Yoon YC. The outcome of ultrasound-guided needle decompression and steroid injection in calcific tendinitis. J Shoulder Elbow Surg. 2010 Jun;19(4):596-600. doi: 10.1016/j.jse.2009.09.002. Epub 2009 Dec 2. PMID 19959377
- [Background] Aina R, Cardinal E, Bureau NJ, Aubin B, Brassard P. Calcific shoulder tendinitis: treatment with modified US-guided fine-needle technique. Radiology. 2001 Nov;221(2):455-61. doi: 10.1148/radiol.2212000830. PMID 11687690
- [Background] Sconfienza LM, Bandirali M, Serafini G, Lacelli F, Aliprandi A, Di Leo G, Sardanelli F. Rotator cuff calcific tendinitis: does warm saline solution improve the short-term outcome of double-needle US-guided treatment? Radiology. 2012 Feb;262(2):560-6. doi: 10.1148/radiol.11111157. Epub 2011 Dec 5. PMID 22143923
- [Background] Guyatt GH, Oxman AD, Vist GE, Kunz R, Falck-Ytter Y, Alonso-Coello P, Schunemann HJ; GRADE Working Group. GRADE: an emerging consensus on rating quality of evidence and strength of recommendations. BMJ. 2008 Apr 26;336(7650):924-6. doi: 10.1136/bmj.39489.470347.AD. PMID 18436948
- [Background] Cohen J. Weighted kappa: nominal scale agreement with provision for scaled disagreement or partial credit. Psychol Bull. 1968 Oct;70(4):213-20. doi: 10.1037/h0026256. No abstract available. PMID 19673146
- [Background] Viera AJ, Garrett JM. Understanding interobserver agreement: the kappa statistic. Fam Med. 2005 May;37(5):360-3. PMID 15883903
- [Background] Zhu J, Jiang Y, Hu Y, Xing C, Hu B. Evaluating the long-term effect of ultrasound-guided needle puncture without aspiration on calcifying supraspinatus tendinitis. Adv Ther. 2008 Nov;25(11):1229-34. doi: 10.1007/s12325-008-0115-x. PMID 18998062
- [Background] Chiou HJ, Chou YH, Wu JJ, Huang TF, Ma HL, Hsu CC, Chang CY. The role of high-resolution ultrasonography in management of calcific tendonitis of the rotator cuff. Ultrasound Med Biol. 2001 Jun;27(6):735-43. doi: 10.1016/s0301-5629(01)00353-2. PMID 11516532
- [Background] De Zordo T, Ahmad N, Odegaard F, Girtler MT, Jaschke W, Klauser AS, Chhem RK, Romagnoli C. US-guided therapy of calcific tendinopathy: clinical and radiological outcome assessment in shoulder and non-shoulder tendons. Ultraschall Med. 2011 Jan;32 Suppl 1:S117-23. doi: 10.1055/s-0029-1245333. Epub 2010 Apr 22. PMID 20414859
- [Background] Farin PU, Rasanen H, Jaroma H, Harju A. Rotator cuff calcifications: treatment with ultrasound-guided percutaneous needle aspiration and lavage. Skeletal Radiol. 1996 Aug;25(6):551-4. doi: 10.1007/s002560050133. PMID 8865489
- [Background] Oliva F, Via AG, Maffulli N. Physiopathology of intratendinous calcific deposition. BMC Med. 2012 Aug 23;10:95. doi: 10.1186/1741-7015-10-95. PMID 22917025
- [Background] Ogon P, Suedkamp NP, Jaeger M, Izadpanah K, Koestler W, Maier D. Prognostic factors in nonoperative therapy for chronic symptomatic calcific tendinitis of the shoulder. Arthritis Rheum. 2009 Oct;60(10):2978-84. doi: 10.1002/art.24845. PMID 19790063
- [Background] Vignesh KN, McDowall A, Simunovic N, Bhandari M, Choudur HN. Efficacy of ultrasound-guided percutaneous needle treatment of calcific tendinitis. AJR Am J Roentgenol. 2015 Jan;204(1):148-52. doi: 10.2214/AJR.13.11935. PMID 25539250
- [Result] Speed CA, Hazleman BL. Calcific tendinitis of the shoulder. N Engl J Med. 1999 May 20;340(20):1582-4. doi: 10.1056/NEJM199905203402011. No abstract available. PMID 10332023
- [Result] Serafini G, Sconfienza LM, Lacelli F, Silvestri E, Aliprandi A, Sardanelli F. Rotator cuff calcific tendonitis: short-term and 10-year outcomes after two-needle us-guided percutaneous treatment--nonrandomized controlled trial. Radiology. 2009 Jul;252(1):157-64. doi: 10.1148/radiol.2521081816. PMID 19561254